CLINICAL TRIAL: NCT00938912
Title: An Open-Label Study To Determine Safety, Tolerability And Efficacy Of Long -Term Oral Lacosamide (LCM) As Adjunctive Therapy In Children With Epilepsy
Brief Title: An Open-Label Study to Determine Safety , Tolerability, and Efficacy of Oral Lacosamide in Children With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP848; 2011-001559-35 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Results first posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2021-12

CONDITIONS: Epilepsy
Keywords: Lacosamide (VIMPAT)
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (Experimental): Subjects and their caregivers may chose to receive Lacosamide oral solution (syrup) or Lacosamide tablets. The maximum duration of LCM administration will be approximately 2 years.
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Lacosamide oral solution (syrup): Total daily dose between 2 mg/kg/day (1 mg/kg bid) to 12 mg/kg/day (6 mg/kg bid)
  Other Names: Vimpat®
Drug: Lacosamide — Lacosamide tablets: Total daily dose between 100 mg (50mg bid) - 600mg (300 mg bid).
  The maximum permissible dose of LCM will be 12 mg/kg/day or 600 mg/day.
  Other Names: Vimpat®

SUMMARY:
SP848 is an open-label study to evaluate long-term safety, tolerability, and efficacy in children with epilepsy treated with Lacosamide (LCM) oral solution (syrup) or LCM tablets as adjunctive therapy.

DETAILED DESCRIPTION:
SP848 is an open-label study to evaluate long-term safety, tolerability, and efficacy in children with epilepsy treated with Lacosamide (LCM) oral solution (syrup) or LCM tablets as adjunctive therapy. In addition, the study is designed to provide continued availability of LCM to subjects who have completed the SP847 (NCT00938431) study and to subjects who have discontinued from SP847 (NCT00938431) and who, in the investigator's opinion, would benefit from long-term administration of LCM.

SP848 will be open to subjects who have participated in other LCM pediatric clinical studies in epilepsy and will also be open to up to 100 subjects enrolling directly into SP848. Permissible LCM doses in SP848 are between 2-12 mg/kg/day (oral solution [syrup]) or the corresponding tablet dose up to a maximum dose of 600 mg/day.

Subjects enrolled in SP848 have the option of remaining on the oral solution formulation of LCM or switching to the commercial tablet formulation, if feasible.

ELIGIBILITY:
Inclusion Criteria:

* A signed informed consent form has been obtained from the parent/legal guardian and assent has been obtained from the subject, as required
* Subject and caregiver (which may be a parent, legal guardian, or other delegated caregiver) are willing and able to comply with all study requirements, including maintaining a daily seizure diary

Subjects who have participated in SP847 or other lacosamide (LCM) pediatric clinical studies in epilepsy must fulfill the following inclusion criteria:

* Subject has completed SP847 (or the subject discontinued SP847 due to a dose reduction or status epilepticus) for the treatment of uncontrolled partial-onset seizures, or subject has participated in other LCM pediatric clinical studies in epilepsy
* Subject is expected to benefit from participation, in the opinion of the investigator

Subjects who enroll directly into SP848 without previous participation in a LCM clinical study must fulfill the following inclusion criteria:

* Subject is >=4 years to <=17 years of age
* Subject has a diagnosis of epilepsy with partial-onset seizures
* Subject has been observed to have uncontrolled partial-onset seizures after an adequate course of treatment (in the opinion of the investigator) with at least 2 Antiepileptic Drugs (AEDs) (concurrently or sequentially)
* Subject has been observed to have at least 2 countable seizures in the 4 week period prior to Screening
* Subject is on a stable dosage regimen of 1 to 3 AEDs
* Subject is an acceptable candidate for venipuncture

Exclusion Criteria:

* Subject is receiving any investigational drugs or using any experimental devices in addition to Lacosamide (LCM)
* Subject >= 6 years of age has a lifetime history of suicide attempt, or has suicidal ideation in the past 6 months

Subjects who have participated in SP847 or other LCM pediatric clinical studies in epilepsy are not permitted to enroll in the study if any of the following criteria are met:

* Subject meets either of the following:

  1. Withdrawal criteria for the primary study (with the exception of subjects who discontinued due to a dose reduction or status epilepticus). For subjects entering from EP0060, if the subject (or legal guardian) withdraws consent solely due to route of LCM administration (iv) or if the subject requires more than 10 iv LCM infusions, the subject may be allowed to participant in SP848 after discussion with and agreement from the Medical Monitor
  2. Ongoing serious Adverse Event (SAE)

     Subjects who enroll directly into SP848 without previous participation in a LCM clinical study are not permitted to enroll in the study if any of the following criteria are met:
* Subject has ever received LCM
* Subject has any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the subject's ability to participate in this study.
* Subject has a medical condition that could reasonably be expected to interfere with drug absorption, distribution, metabolism, or excretion
* Subject has a known hypersensitivity to any component of the investigational medicinal product
* Subject is a female of childbearing potential and does not practice an acceptable method of contraception for the duration of the study
* Subject has a creatinine clearance less than 30mL/min
* Subject has a clinically relevant ECG abnormality, in the opinion of the principal investigator (ie, second or third degree heart block at rest or a QT prolongation greater than 450ms)
* Subject has hemodynamically significant heart disease (eg, heart failure)
* Subject has an arrhythmic heart condition requiring medical therapy
* Subject has a known history of severe anaphylactic reaction or serious blood dyscrasias
* Subject has nonepileptic events, including psychogenic seizures, that could be confused with seizures. If both epileptic and nonepileptic events are present, epileptic events must be distinguished from nonepileptic phenomena
* Subject has a history of primary generalized epilepsy
* Subject is taking monoamine oxidase inhibitors-A (MAOI-A) or narcotic analgesics.
* Subject has epilepsy secondary to a progressing cerebral disease or any other progressively neurodegenerative disease, such as Rasmussen syndrome
* Subject has a known sodium channelopathy, such as Brugada syndrome
* Subject has >2x upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or >ULN total bilirubin (1.5xULN total bilirubin if known Gilbert's syndrome). If subject has elevations only in total bilirubin that are >ULN and <1.5xULN, fractionate bilirubin to identify possible undiagnosed Gilbert's syndrome (ie, direct bilirubin <35%)

Subjects who were directly enrolled in EP0060 for iv LCM replacement therapy or to initiate LCM treatment are not permitted to enroll in the study if any of the following criteria are met:

- Subjects have previously participated in a long-term, open-label LCM study

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 366 (Actual)
Dates: Start 2009-12-09 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273(UCB)
Locations (69):
- United States (24):
  - Sp848 064, Birmingham, Alabama
  - Sp848 059, Los Angeles, California
  - Sp848 025, Sacramento, California
  - Sp848 002, Washington D.C., District of Columbia
  - Sp848 054, Orlando, Florida
  - Sp848 012, Tampa, Florida
  - Sp848 019, Wellington, Florida
  - Sp848 057, Augusta, Georgia
  - Sp848 063, Saint Paul, Minnesota
  - Sp848 006, Saint Paul, Minnesota
  - Sp848 008, Kansas City, Missouri
  - Sp848 061, Las Vegas, Nevada
  - Sp848 062, Hackensack, New Jersey
  - Sp848 015, New Brunswick, New Jersey
  - Sp848 005, Durham, North Carolina
  - Sp848 053, Akron, Ohio
  - Sp848 068, Cincinnati, Ohio
  - Sp848 001, Philadelphia, Pennsylvania
  - Sp848 016, Pittsburgh, Pennsylvania
  - Sp848 004, Nashville, Tennessee
  - Sp848 026, Austin, Texas
  - Sp848 067, Dallas, Texas
  - Sp848 022, Houston, Texas
  - Sp848 020, Norfolk, Virginia
- Belgium (4):
  - Sp848 201, Brussels
  - Sp848 200, Edegem
  - Sp848 203, Ghent
  - Sp848 202, Leuven
- China (7):
  - Sp848 950, Beijing
  - Sp848 953, Changchun
  - Sp848 951, Chongqing
  - Sp848 955, Hanzhou
  - Sp848 956, Nanchang
  - Sp848 952, Shanghai
  - Sp848 954, Shenzhen
- France (2):
  - Sp848 309, Paris
  - Sp848 304, Strasbourg
- Sp848 403, Kork, Germany
- Hungary (5):
  - Sp848 701, Budapest
  - Sp848 702, Budapest
  - Sp848 703, Budapest
  - Sp848 704, Budapest
  - Sp848 705, Debrecen
- Italy (2):
  - Sp848 503, Messina
  - Sp848 502, Verona
- Japan (9):
  - Sp848 257, Fukuoka
  - Sp848 256, Hamamatsu
  - Sp848 255, Kodaira
  - Sp848 253, Kōshi
  - Sp848 252, Niigata
  - Sp848 258, Okayama
  - Sp848 254, Osaka
  - Sp848 259, Osaka
  - Sp848 251, Shizuoka
- Mexico (3):
  - Sp848 101, Culiacán
  - Sp848 104, Guadalajara
  - Sp848 103, San Luis Potosí City
- Poland (5):
  - Sp848 803, Bialystok
  - Sp848 807, Katowice
  - Sp848 804, Kielce
  - Sp848 801, Krakow
  - Sp848 805, Lublin
- Ukraine (7):
  - Sp848 224, Dnipro
  - Sp848 225, Dnipro
  - Sp848 220, Ivano-Frankivsk
  - Sp848 221, Kiev
  - Sp848 222, Kiev
  - Sp848 226, Kiev
  - Sp848 223, Vinnytsia

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in December 2009 and concluded in May 2021. Eligible study participants were allowed to roll over from study SP0847 (NCT00938431), SP0966 (NCT01969851) and EP0060 (NCT02710890) and eligible study participants were also allowed to directly enroll into the study.
Pre-assignment Details: Total 366 participants were enrolled. Among 366, 365 participants received treatment. One participant was enrolled, but did not receive treatment prior to discontinuing due to ineligibility.
Groups:
- Lacosamide (All Participants): Participants aged greater than or equal to (≥1) month received either lacosamide (LCM) 2-12 milligrams/kilograms/day (mg/kg/day) (oral solution) or 100-600 mg/day (tablet) at a level to optimize tolerability and seizure control (maximum dose of 12 mg/kg/day or 600 mg/day based on body weight, whichever was lower) for approximately 2 years.
Period: Overall Study
Arm/Group | Lacosamide (All Participants)
Started | 365
Completed | 254
Not Completed | 111
Not completed — Withdrawal by Subject | 28
Not completed — Lost to Follow-up | 4
Not completed — Lack of Efficacy | 43
Not completed — Adverse event, non-fatal | 24
Not completed — Adverse event, fatal | 1
Not completed — Participant self adjusted antiepileptic medication | 1
Not completed — Participant had a creatinine clearance less than 30 mL/min | 1
Not completed — Participant needed prohibit medication | 1
Not completed — Participant was scheduled for lobal resection | 1
Not completed — Did not meet Eligibility criteria | 1
Not completed — Participant relocated not related to AE | 1
Not completed — Participant moved to another city | 1
Not completed — Participant experienced break through seizures | 1
Not completed — No longer wished to participate in the study | 1
Not completed — Protocol Deviation | 2

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the SS which consisted of all enrolled study participants who took at least 1 dose of LCM in this study.
Groups:
- Lacosamide (All Participants): Participants aged ≥1 month received either LCM 2-12 mg/kg/day (oral solution) or 100-600 mg/day (tablet) at a level to optimize tolerability and seizure control (maximum dose of 12 mg/kg/day or 600 mg/day based on body weight, whichever was lower) for approximately 2 years.
Arm/Group | Lacosamide (All Participants)
Number analyzed (Participants) | 365
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 365
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.28 (4.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173
  Male | 192
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan native | 1
  Asian | 111
  Black | 26
  White | 201
  Other/Mixed | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With At Least One Treatment-Emergent Adverse Event (TEAE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation study participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. TEAEs were defined as those events which started on or after the date of first SP848 LCM administration and occurred within 30 days after last dose of LCM, or whose severity worsened on or after the date of first SP848 LCM administration.
Time Frame: From Baseline to End of Safety Follow-Up (up to 4.3 years)
Population: The Safety Set (SS) consisted of all enrolled study participants who took at least 1 dose of LCM in this study.
Measure: Count of Participants; unit: Participants
Groups:
- Lacosamide (All Participants) (SS): Participants aged ≥1 month received either LCM 2-12 mg/kg/day (oral solution) or 100-600 mg/day (tablet) at a level to optimize tolerability and seizure control (maximum dose of 12 mg/kg/day or 600 mg/day based on body weight, whichever was lower) for approximately 2 years. Participants formed the Safety Set (SS) which included all enrolled study participants who took at least 1 dose of LCM in this study.
Arm/Group | Lacosamide (All Participants) (SS)
Number analyzed (Participants) | 365
Participants | 336

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: SAE was any untoward medical occurrence that at any dose resulted in death, is life-threatening, required in participant hospitalization or prolongation of existing hospitalization, is a congenital anomaly or birth defect, is an infection that requires treatment with parenteral antibiotics, other important medical events which based on medical or scientific judgement may jeopardize the participants, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Baseline to End of Safety Follow-Up (up to 4.3 years)
Population: The SS consisted of all enrolled study participants who took at least 1 dose of LCM in this study.
Measure: Count of Participants; unit: Participants
Groups:
- Lacosamide (All Participants) (SS): Participants aged ≥1 month received either LCM 2-12 mg/kg/day (oral solution) or 100-600 mg/day (tablet) at a level to optimize tolerability and seizure control (maximum dose of 12 mg/kg/day or 600 mg/day based on body weight, whichever was lower) for approximately 2 years. Participants formed the SS which included all enrolled study participants who took at least 1 dose of LCM in this study.
Arm/Group | Lacosamide (All Participants) (SS)
Number analyzed (Participants) | 365
Participants | 82

3. Primary Outcome: Number of Participants That Withdraw Due to a Treatment-Emergent Adverse Event
Description: TEAEs were defined as those events which started on or after the date of first SP848 LCM administration and occurred within 30 days after last dose of LCM, or whose severity worsened on or after the date of first SP848 LCM administration.
Time Frame: From Baseline to End of Safety Follow-Up (up to 4.3 years)
Population: The SS consisted of all enrolled study participants who took at least 1 dose of LCM in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide (All Participants) (SS)
Number analyzed (Participants) | 365
Participants | 27

4. Secondary Outcome: Percent Change From Baseline in 28 Day Partial-onset Seizure Frequency to the End of the Treatment Period
Description: Percent change in seizure frequency per 28 days (PCH) from the Baseline value (B) to Treatment Period interval (T) was defined as:PCH = [(SFT - SFB)/SFB] x 100 where, SFT corresponded to seizure frequency during Treatment Period for relative interval in open-label study and SFB corresponded to Baseline seizure frequency. For both periods, the frequency was standardized to the number of seizures per 28 days. For rollover participants, the Baseline values from the previous pediatric studies were designated as Baseline values in SP848. The Baseline value for seizure counts for directly enrolled participants were taken from the historical seizure count case report form/electronic case report form (CRF/eCRF) module in combination with the seizure diary data collected from the date of the Screening Visit to the day prior to the date of first dose of LCM. Participants from EP0060 RxL enrollment group had no baseline data due to taking oral LCM prior to EP0060.
Time Frame: From Baseline to End of Treatment Period (up to 4.2 years)
Population: The Full Analysis Set (FAS) consisted of all study participants in the SS who had at least 1 completed post-Baseline seizure diary. Here, number of participants analyzed included those participants who were evaluable for the assessment.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Lacosamide (All Participants) (FAS): Participants aged ≥1 month received either LCM 2-12 mg/kg/day (oral solution) or 100-600 mg/day (tablet) at a level to optimize tolerability and seizure control (maximum dose of 12 mg/kg/day or 600 mg/day based on body weight, whichever was lower) for approximately 2 years. Participants formed the Full Analysis Set (FAS) which included all study participants in the SS who had at least 1 completed post-Baseline seizure diary.
Arm/Group | Lacosamide (All Participants) (FAS)
Number analyzed (Participants) | 308
percent change | -24.13 (112.08)

5. Secondary Outcome: Percentage of Participants With ≥50% Reduction in 28-day Partial-onset Seizure Frequency
Description: A 50% responder is a participant experiencing a ≥50% reduction in partial-onset seizure frequency per 28 days from Baseline to end of the specified time interval, otherwise a participant is a non-responder. For rollover participants, the Baseline values from the previous pediatric studies were designated as Baseline values in SP848. The Baseline value for seizure counts for directly enrolled participants were taken from the historical seizure count CRF/eCRF module in combination with the seizure diary data collected from the date of the Screening Visit to the day prior to the date of first dose of LCM. Participants from EP0060 RxL enrollment group had no baseline data due to taking oral LCM prior to EP0060.
Time Frame: From Baseline to End of Treatment Period (up to 4.2 years)
Population: The FAS consisted of all study participants in the SS who had at least 1 completed post-Baseline seizure diary. Here, number of participants analyzed included those participants who were evaluable for the assessment.
Measure: Number; unit: percentage of participants
Groups:
- Lacosamide (All Participants) (FAS): Participants aged ≥1 month received either LCM 2-12 mg/kg/day (oral solution) or 100-600 mg/day (tablet) at a level to optimize tolerability and seizure control (maximum dose of 12 mg/kg/day or 600 mg/day based on body weight, whichever was lower) for approximately 2 years. Participants formed the FAS which included all study participants in the SS who had at least 1 completed post-Baseline seizure diary.
Arm/Group | Lacosamide (All Participants) (FAS)
Number analyzed (Participants) | 308
percentage of participants | 53.6

6. Secondary Outcome: Percentage of Participants With ≥75% Reduction in 28-day Partial-onset Seizure Frequency
Description: A 75% responder is a participant experiencing a ≥75% reduction in partial-onset seizure frequency per 28 days from Baseline to end of the specified time interval, otherwise a participant is a non-responder. For rollover participants, the Baseline values from the previous pediatric studies were designated as Baseline values in SP848. The Baseline value for seizure counts for directly enrolled participants were taken from the historical seizure count CRF/eCRF module in combination with the seizure diary data collected from the date of the Screening Visit to the day prior to the date of first dose of LCM. Participants from EP0060 RxL enrollment group had no baseline data due to taking oral LCM prior to EP0060.
Time Frame: From Baseline to End of Treatment Period (up to 4.2 years)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide (All Participants) (FAS)
Number analyzed (Participants) | 308
percentage of participants | 40.3

7. Secondary Outcome: Number of Seizure Days Per 28 Days for Participants With Generalized Seizures
Description: A seizure day was defined as a day where any type of seizure was reported in the seizure diary and seizures were assessed. Days in the seizure diary which were marked as "not done" on the CRF/eCRF were not counted as seizure-free days.
Time Frame: Weeks 4, 8, 12, 20, 28, 36, 44, 52, 60, 72, 84 and 96
Population: The FAS consisted of all study participants in the SS who had at least 1 completed post-Baseline seizure diary. Here, number of participants analyzed included those participants who were evaluable for the assessment and number analyzed signifies participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: seizure days per 28 days
Arm/Group | Lacosamide (All Participants) (FAS)
Number analyzed (Participants) | 47
seizure days per 28 days
  Week 4 | 14.59 (11.94)
  Week 8: number analyzed (Participants) | 46
  Week 8 | 14.83 (12.24)
  Week 12: number analyzed (Participants) | 46
  Week 12 | 13.68 (12.62)
  Week 20: number analyzed (Participants) | 46
  Week 20 | 12.57 (12.58)
  Week 28: number analyzed (Participants) | 43
  Week 28 | 13.10 (12.63)
  Week 36: number analyzed (Participants) | 43
  Week 36 | 11.43 (11.93)
  Week 44: number analyzed (Participants) | 40
  Week 44 | 9.24 (11.23)
  Week 52: number analyzed (Participants) | 41
  Week 52 | 10.48 (11.68)
  Week 60: number analyzed (Participants) | 39
  Week 60 | 10.31 (11.84)
  Week 72: number analyzed (Participants) | 39
  Week 72 | 11.15 (12.10)
  Week 84: number analyzed (Participants) | 38
  Week 84 | 11.87 (12.45)
  Week 96: number analyzed (Participants) | 37
  Week 96 | 10.73 (11.77)

8. Secondary Outcome: Percentage of Participants Who Achieved a Seizure-free Status
Description: Study participants were considered seizure-free for a given period if they completed the period, reported zero seizures during the period, and had no more than 10% of days in the period for which seizure data were not available (ie, "not done" was noted on the Seizure Frequency CRF/eCRF module).
Time Frame: From Baseline to End of Treatment Period (up to 4.2 years)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide (All Participants) (FAS)
Number analyzed (Participants) | 323
percentage of participants | 7.4

ADVERSE EVENTS:
Time Frame: From Baseline to End of Safety Follow-Up (up to 4.3 years)
Description: TEAEs were defined as those events which started on or after the date of first SP848 LCM administration and occurred within 30 days after last dose of LCM, or whose severity worsened on or after the date of first SP848 LCM administration.
Arm/Group | Lacosamide (All Participants) (SS)
All-Cause Mortality (participants affected / at risk) | 1/365
Serious Adverse Events (participants affected / at risk) | 82/365
Other Adverse Events (participants affected / at risk) | 291/365
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (All Participants) (SS) (N=365)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cyanosis (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (19)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Intussusception (Gastrointestinal disorders) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Traumatic tooth displacement (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 4 (5)
Adverse drug reaction (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Bronchitis (Infections and infestations) | 4 (4)
Bronchopneumonia (Infections and infestations) | 3 (3)
Gastroenteritis (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Otitis media (Infections and infestations) | 2 (2)
Tonsillitis (Infections and infestations) | 2 (3)
Acute tonsillitis (Infections and infestations) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Erythema infectiosum (Infections and infestations) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (2)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1)
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Atlantoaxial instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Astrocytoma, low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Convulsion (Nervous system disorders) | 21 (29)
Status epilepticus (Nervous system disorders) | 11 (16)
Epilepsy (Nervous system disorders) | 6 (6)
Complex partial seizures (Nervous system disorders) | 5 (6)
Partial seizures with secondary generalisation (Nervous system disorders) | 4 (12)
Partial seizures (Nervous system disorders) | 3 (3)
Seizure cluster (Nervous system disorders) | 3 (5)
Headache (Nervous system disorders) | 2 (2)
Altered state of consciousness (Nervous system disorders) | 1 (1)
Clonic convulsion (Nervous system disorders) | 1 (1)
Encephalitis autoimmune (Nervous system disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Neurotoxicity (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Psychomotor skills impaired (Nervous system disorders) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1)
Simple partial seizures (Nervous system disorders) | 1 (2)
Somnolence (Nervous system disorders) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (5)
Affective disorder (Psychiatric disorders) | 1 (2)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (2)
Hallucination, visual (Psychiatric disorders) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (All Participants) (SS) (N=365)
Vomiting (Gastrointestinal disorders) | 77 (149)
Diarrhoea (Gastrointestinal disorders) | 40 (52)
Constipation (Gastrointestinal disorders) | 25 (34)
Nausea (Gastrointestinal disorders) | 25 (35)
Abdominal pain (Gastrointestinal disorders) | 21 (32)
Abdominal pain upper (Gastrointestinal disorders) | 19 (29)
Pyrexia (General disorders) | 80 (126)
Fatigue (General disorders) | 21 (31)
Nasopharyngitis (Infections and infestations) | 91 (253)
Upper respiratory tract infection (Infections and infestations) | 86 (167)
Pharyngitis (Infections and infestations) | 37 (48)
Gastroenteritis (Infections and infestations) | 29 (35)
Influenza (Infections and infestations) | 29 (38)
Bronchitis (Infections and infestations) | 26 (40)
Viral infection (Infections and infestations) | 21 (36)
Sinusitis (Infections and infestations) | 20 (29)
Urinary tract infection (Infections and infestations) | 20 (24)
Ear infection (Infections and infestations) | 19 (27)
Contusion (Injury, poisoning and procedural complications) | 25 (55)
Decreased appetite (Metabolism and nutrition disorders) | 26 (28)
Somnolence (Nervous system disorders) | 74 (100)
Dizziness (Nervous system disorders) | 69 (114)
Headache (Nervous system disorders) | 45 (97)
Tremor (Nervous system disorders) | 21 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 36 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT00938912/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT00938912/SAP_001.pdf